CLINICAL TRIAL: NCT00719680
Title: A Multicenter Extension Study of the Efficacy, Tolerability, and Safety of Immune Globulin Subcutaneous (Human) IgPro20 in Subjects With Primary Immunodeficiency (PID)
Brief Title: Extension Study of Subcutaneous Immunoglobulin Human in Patients With Primary Immunodeficiency (PID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_3001; 1473 (Other: CSL Behring)
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2012-12

CONDITIONS: Primary Immune Deficiency
Keywords: CVID; XLA
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Hizentra; Immunoglobulin G; Proline

ARMS (1):
- IgPro20 (Experimental): The IgPro20 dose will be the same as in the previous pivotal study ZLB04_009CR (NCT00419341) infused subcutaneously weekly or twice a week (in the latter case, half of a weekly dose will be used)
  Interventions: Biological: IgPro20

INTERVENTIONS:
Biological: IgPro20
  Other Names: IgG with Proline

SUMMARY:
The purpose of this study is to determine whether a long-term use of a new human immunoglobulin G with proline (IgPro) is safe and effective in the treatment of primary immunodeficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with primary humoral immunodeficiency who have participated in the study ZLB04_009CR (NCT00419341), namely with a diagnosis of Common Variable Immunodeficiency (CVID) as defined by PAGID (Pan-American Group for Immunodeficiency) and ESID (European Society for Immunodeficiencies) or X-linked Agammaglobulinemia (XLA) as defined by PAGID and ESID
* Women of childbearing potential must be using and agree to continue using medically approved contraception and must have a negative pregnancy test at screening
* Written informed consent

Exclusion Criteria:

* Ongoing serious bacterial infection at the time of screening
* Malignancies of lymphoid cells such as lymphocytic leukemia, Non-Hodgkin's lymphoma, and immunodeficiency with thymoma
* Hypoalbuminemia, protein-losing enteropathies, and any proteinuria (defined by total urine protein concentration > 0.2 g/L)
* Other significant medical conditions that could increase the risk to the patient
* Females who are pregnant, breast-feeding or planning a pregnancy during the course of the study
* A positive result at screening on any of the following viral markers: Human immunodeficiency virus (HIV), Hepatitis C virus (HCV) or Hepatitis B virus (HBV)
* Aspartate aminotransferase (ASAT) or Alanine aminotransferase (ALAT) concentration > 2.5 times Upper Normal Limit (UNL) at Completion Visit of study ZLB04_009CR (NCT00419341)
* Creatinine concentration > 1.5 times UNL at Completion Visit of study ZLB04_009CR (NCT00419341)
* Participation in a study with an investigational product other than IgPro20 within 3 months prior to enrollment
* Evidence of uncooperative attitude
* Any condition that is likely to interfere with evaluation of the study drug or satisfactory conduct of the trial
* Subjects who are employees at the investigational site, relatives or spouse of the investigator

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (4):
- United States (4):
  - Contact CSL Behring for facility details, Centennial, Colorado
  - Contact CSL Behring for facility details, North Palm Beach, Florida
  - Contact CSL Behring for facility details, Indianapolis, Indiana
  - Contact CSL Behring for facility details, Dallas, Texas

REFERENCES:
- [Result] Jolles S, Borte M, Nelson RP Jr, Rojavin M, Bexon M, Lawo JP, Wasserman RL. Long-term efficacy, safety, and tolerability of Hizentra(R) for treatment of primary immunodeficiency disease. Clin Immunol. 2014 Feb;150(2):161-9. doi: 10.1016/j.clim.2013.10.008. Epub 2013 Oct 26. PMID 24412910

RESULTS

PARTICIPANT FLOW:
Groups:
- IgPro20: A liquid formulation of normal human IgG at a concentration of 20%. IgPro20 was administered as a subcutaneous infusion weekly or twice weekly, depending on the investigator's judgment and the subject's preference.
Period: Overall Study
Arm/Group | IgPro20
Started | 21
Completed | 16
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (18.53)
Age, Customized [Number; unit: participants]
  >= 2 to < 12 years | 1
  >= 12 to < 16 years | 1
  >= 16 to < 65 years | 16
  >= 65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Serious Bacterial Infection (Intention-to-Treat Population)
Description: The annualized rate was based on the total number of infections and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
  Acute serious bacterial infections included pneumonia, bacteremia/septicemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The Intention-to-Treat (ITT) population comprised all subjects treated with study medication during any study period.
Measure: Number; unit: infections per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Subject Study Days) | 11950
infections per subject year | 0.06

2. Secondary Outcome: Annualized Rate of Any Infection
Description: The annualized rate was based on the total number of infections and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Number; unit: infections per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Subject Study Days) | 11950
infections per subject year | 2.38

3. Primary Outcome: Annualized Rate of Serious Bacterial Infection (Per-Protocol Efficacy Population)
Description: as for outcome 1
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The Per-Protocol Efficacy population comprised all subjects who completed at least 48 weeks of the efficacy period that started with the first IgPro20 dose in this study.
Measure: Number; unit: infections per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 18
Number analyzed (Subject Study Days) | 11037
infections per subject year | 0.03

4. Secondary Outcome: Trough Levels of Total Immunoglobulin G (IgG) Serum Concentrations
Description: Mean of individual median total IgG trough concentration.
Time Frame: Before infusion at Weeks 1, 24, 48, 72, and 96
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | IgPro20
Number analyzed (Participants) | 21
g/L | 11.98 (3.65)

5. Secondary Outcome: Number of Days Out of Work / School / Kindergarten / Day Care or Inability to Perform Normal Activities Due to Infection
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
days | 6.67 (13.49)

6. Secondary Outcome: Annualized Rate of Days Out of Work / School / Kindergarten / Day Care or Inability to Perform Normal Activities Due to Infection
Description: The annualized rate was based on the total number of days out of work / school / kindergarten / day care or inability to perform normal activities due to infection, and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Subject Study Days) | 11950
days per subject year | 4.28

7. Secondary Outcome: Number of Days of Hospitalization Due to Infection
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
days | 0.857 (2.726)

8. Secondary Outcome: Annualized Rate of Hospitalization Due to Infection
Description: The annualized rate was based on the total number of days of hospitalization due to infection and the total number of subject study days for all subjects in the specified analysis population and adjusted to 365 days.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Study Days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Subject Study Days) | 11950
days per subject year | 0.55

9. Secondary Outcome: Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Annualized rate of days with antibiotics for infection prophylaxis and treatment.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The ITT population comprised all subjects treated with study medication during any study period.
Measure: Number; unit: days per subject year
Units Other Than Participants: Subject Exposure Days
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Subject Exposure Days) | 11950
days per subject year | 83.87 [5 to 673]

10. Secondary Outcome: Rate of All AEs by Relatedness and Severity
Description: The rate of AEs was the number of AEs over the number of infusions administered.
  At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The All-Treated (AT) safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Infusions) | 1735
AEs per infusion
  All | 0.661
  Unrelated | 0.137
  At least possibly related | 0.524
  Mild | 0.575
  Moderate | 0.076
  Severe | 0.010

11. Secondary Outcome: Relatedness and Severity of All AEs (Percentage of Total AEs)
Description: At least possibly related AEs included possibly related AEs, probably related AEs, and related AEs.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: percentage of total AEs
Units Other Than Participants: AEs
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (AEs) | 1147
percentage of total AEs
  Unrelated | 20.7
  At least possibly related | 79.3
  Mild | 87.0
  Moderate | 11.5
  Severe | 1.5

12. Secondary Outcome: Number of Subjects With Any Temporally Associated Adverse Event (AE) Within 24 or 72 Hours After an Infusion
Description: AEs were considered temporally associated if they occurred between the start of infusion and within 24 or 72 hours after the end of infusion.
Time Frame: Within 24 or 72 hours after each infusion
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 21
participants
  AEs within 24 hours | 21
  AEs within 72 hours | 21

13. Secondary Outcome: Rate of Temporally Associated AEs Within 24 or 72 Hours of an Infusion
Description: The rate of AEs was the number of AEs over the number of infusions administered.
  AEs were considered temporally associated if they occurred between the start of infusion and within 24 or 72 hours after the end of infusion.
Time Frame: Within 24 or 72 hours after each infusion
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro20
Number analyzed (Participants) | 21
Number analyzed (Infusions) | 1735
AEs per infusion
  AEs within 24 hours | 0.322
  AEs within 72 hours | 0.575

14. Secondary Outcome: Number of Subjects Reporting Mild, Moderate, or Severe Local AEs
Description: In addition to the standard MedDRA System Organ Class (SOC) AE assignments, the category of 'local reactions' was defined to provide the possibility for a combined analysis of local reactions and included AEs of infusion site oedema, infusion site reaction, injection site pain, injection site rash, and injection site reaction.
  Mild AE: Did not interfere with routine activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
Time Frame: For the duration of the study, up to approximately 104 weeks
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 21
participants
  Total | 19
  Mild | 16
  Moderate | 3
  Severe | 0

15. Secondary Outcome: Number of Subjects With Clinically Significant Changes From Baseline to the Completion Visit in Vital Signs
Description: Vital signs included blood pressure (systolic and diastolic), heart rate, and body temperature.
Time Frame: At weeks 1, 12, 24, 36, 48, 60, 72, 84, and 96
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 21
participants | 0

16. Secondary Outcome: Number of Subjects With Clinically Significant Changes From Baseline to the Completion Visit in Routine Laboratory Parameters
Description: Routine laboratory parameters included hematology, blood chemistry, and urinalysis parameters.
Time Frame: At Week 1, and study completion (approximately 104 weeks)
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 21
participants | 0

17. Secondary Outcome: Number of Subjects With Clinically Significant Changes From Baseline to the Completion Visit in Viral Safety Markers
Description: Viral safety markers included human immunodeficiency virus (HIV)-1, HIV-2, hepatitis A virus (HAV), HBV, HCV, and parvovirus B19.
Time Frame: At Week 1, and study completion (approximately 104 weeks)
Population: The AT safety population comprised all subjects treated with the study medication during any study period.
Measure: Number; unit: participants
Arm/Group | IgPro20
Number analyzed (Participants) | 21
participants | 0

ADVERSE EVENTS:
Time Frame: From the time of informed consent until study completion, up to approximately 121 weeks
Description: The All-Treated (AT) safety population comprised all subjects treated with the study medication during any study period
Arm/Group | IgPro20
Serious Adverse Events (participants affected / at risk) | 4/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=21)
Cellulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (N=21)
Injection site reaction (General disorders) | 10 (248)
Infusion site reaction (General disorders) | 9 (614)
Nasopharyngitis (Infections and infestations) | 7 (10)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Fatigue (General disorders) | 5 (33)
Influenza-like illness (General disorders) | 4 (7)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (10)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Headache (Nervous system disorders) | 3 (10)
Abdominal pain upper (Gastrointestinal disorders) | 2 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Chest pain (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Depression (Psychiatric disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (4)
Injection site pain (General disorders) | 2 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (4)
Migraine (Nervous system disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3)
Pyrexia (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 5 (7)
Clostridial infection (Infections and infestations) | 2 (3)
Pharyngitis (Infections and infestations) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 6 (6)
Viral infection (Infections and infestations) | 2 (4)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 14 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and requests that reports based on single-site data not precede the primary publication of the entire clinical trial.